CLINICAL TRIAL: NCT06544525
Title: Is Conditioned Pain Modulation Predictive of Clinical Improvement in Patients With Chronic Low Back Pain?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kyle R. Petrey, Orthopedic and Manual Physical Therapy Fellow, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.2024.070
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: low back pain; physical therapy; conditioned pain modulation; temporal summation
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This study will be a quasi-experimental, one-group repeated measures design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- chronic low back pain (Experimental): Age 18-64 years with low back pain duration greater than 3 months.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy — The intervention will be physical therapy standard of care.

SUMMARY:
Conditioned pain modulation (CPM) a measure of the effectiveness of the descending pain pathway and therefore a measure of the body's ability to perform endogenous analgesia. In subjects with normal function of the descending pain pathway, the net-effect during CPM testing is anti-nociceptive, or inhibition of the ascending pain pathway. In those with impaired descending pain pathway function, the response to CPM testing is pro-nociceptive, indicating that the body is unable to inhibit the pain signal, or may even amplify it. There is literature that supports the presence of impaired CPM, and therefore impaired descending pain pathway function, in numerus chronic pain conditions, including low back pain. Impaired descending pain pathway function may be contributing to this chronic pain presentation. This study will give us information on whether a typical physical therapy plan of care is able to improve impaired CPM, and if CPM values are predictive of improvement in physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* DEERS eligible
* English speaking
* Age 18-64 years
* ODI baseline ≥25%
* NPRS baseline ≥3/10
* Low back pain symptoms greater than 3 months
* Must be able to commit to at least six weeks of physical therapy interventions

Exclusion Criteria:

* Serious spinal pathology (acute fracture, active cancer, inflammation, inflammatory arthropathy)
* Low back pain symptoms radiating below the knee
* Pregnancy
* Diagnosed neurological disease including traumatic brain injury, multiple sclerosis, chronic regional pain syndrome, and fibromyalgia.
* History spinal surgery
* Currently under litigation related to low back pain
* Currently going through Medical Evaluation Board (MEB)
* Retiring or separating from the military within a year

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Modified Oswestry Disability Index | From enrollment until end of study at 6 weeks.
  The ODI will be the primary outcome for this study. The ODI contains 10 items that assess function and disability (0 = no disability, 100 = maximal disability).

SECONDARY OUTCOMES:
Central Sensitization Inventory | From enrollment until study end at 6 weeks.
  The CSI is a 25-item questionnaire that assesses symptoms common to central sensitization syndromes using a 0-100-point scale, in which 100 indicates a higher level of symptoms common to central sensitization.
Conditioned pain modulation | From enrollment until study end at 6 weeks.
  CPM calculation: It is recommended that CPM response be reported as an absolute value and percent change. The calculation for absolute value is: CPM = PPTpre -PPTconditioning. PPTpre is the testing stimulus conducted before conditioning stimulus application and PPTconditioning is the testing stimulus conducted during conditioning stimulation. This is expressed in kPa. A negative value suggests that CPM is functioning effectively and indicative of an anti-nociceptive profile, while a positive value suggests CPM is impaired and indicative of a pro-nociceptive profile. The second method will be CPM expressed as percent change of the testing stimulus before and during the application of the conditioning stimulus. The equation for percent change is: [(postPPT - prePPT)/prePPT] * 100. CPM will be expressed as continuous ratio data via absolute value and percent change. The absolute value score will be used for the statistical model and will be collected at baseline and follow up.
Temporal Summation | From enrollment until study end at 6 weeks.
  Temporal summation is calculated as follows: VAS10th - VAS1st. A positive number indicates the magnitude of temporal summation of pain. This will be expressed as continuous ratio data and will be collected at baseline and follow up.
Numeric pain rating scale | From enrollment until study end (6 weeks).
  The NPRS is an 11-point numerical pain rating scale used to measure pain. Patients rate pain ranging between 0 (no pain) and 10 (worst pain imaginable).
  This will be measured as the mean of three pain ratings: best pain rating over 24 hours, worst pain rating over 24 hours, and current pain rating.
Global rating of change scale | From enrollment until end of study (6 weeks)
  The GRC utilized in this study is an 11-point scale designed to quantify a patient's improvement or deterioration over time. The GRC will only be completed at discharge (6-weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Petrey, DPT, Principal Investigator — BAMC
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for deidentified data will be considered on a case by case basis.
Supporting Information: Study Protocol
Time Frame: Requests for deidentified data will be considered on a case by case basis.
Access Criteria: Requests for deidentified data will be considered on a case by case basis.